CLINICAL TRIAL: NCT00022997
Title: Studies of Deficits in the Sense of Taste
Brief Title: Study of Taste Deficits
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010230; 01-DC-0230
Record Dates: First submitted 2001-08-17; First posted 2001-08-20 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06-04

CONDITIONS: Taste Disorder; Healthy
Keywords: Phenylthiocarbamide; Phlebotomy; Chemoreceptors; Population Associations; Non-Tasters; Taste; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Taste Disorders

SUMMARY:
This study will explore the genetics of taste and taste deficits. The sense of taste plays a crucial role in food choices, allowing people to identify beneficial foods (those with high caloric value, which are typically sweet) and foods likely to be toxic (usually bitter substances). The loss of sense of taste in older people plays a role in decreased appetite and poor nutrition. Taste deficits may adversely affect people in ways that are not well understood. This study will examine why some people (about one-fourth of all people in the United States) cannot taste a substance called phenylthiocarbamide (PTC). The inability to taste PTC is due to inherited factors that are not yet clear.

Individuals age 18 and older who can taste PTC and individuals who cannot taste PTC may be eligible for this study. Participants will taste a number of liquid solutions until they find one with a clear taste. Then they will taste another group of solutions and decide which ones have that taste and which have no taste. Finally, they will taste a third group of solutions until they find one with a different taste. About 2 tablespoons of blood will be drawn from participants for genetic tests related to the sense of taste.

DETAILED DESCRIPTION:
The primary goal of this study is to identify the underlying cause of deficits in the ability to taste different commonly consumed substances, including the bitter compound phenylthiocarbamide (PTC) as a model. Individuals will be tested to identify those who can and cannot taste PTC, as well as for their ability to taste a variety of sweet, sour, salty, and savory substances. Individuals will have 20 cc of blood drawn to obtain DNA. These DNA samples will then be analyzed for variation in genes whose products are known to be involved in taste perception pathways. Information about individuals DNA sequence variation will then be correlated with their taste phenotype to identify the specific genetic variation that causes phenotypic variation, providing molecular structure-function information in taste sensory pathways.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals age 18 years and older.
* Subjects must be medically healthy, with no cognitive impairment or physical swallowing inability or impairment
* Must be able to provide informed consent
* Must be able to read and understand English.
* NIH employees or staff may participate in this study if they meet the eligibility criteria.

EXCLUSION CRITERIA:

* Cannot be younger than 18 years of age
* Subjects with suspected or known cognitive impairment or physical swallowing inability or impairment
* Subjects who are unable to provide informed consent
* Subjects who are taking any pyschoactive medications or medications that affect their nervous system, such as antidepressants or anti-psychotics.
* Subjects who have known problems with these sense of taste
* Subjects who are currently using tobacco

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2001-08-16; Study Completion 2019-06-04

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Drayna, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Reddy BM, Rao DC. Phenylthiocarbamide taste sensitivity revisited: complete sorting test supports residual family resemblance. Genet Epidemiol. 1989;6(3):413-21. doi: 10.1002/gepi.1370060304. PMID 2753351
- [Background] Adler E, Hoon MA, Mueller KL, Chandrashekar J, Ryba NJ, Zuker CS. A novel family of mammalian taste receptors. Cell. 2000 Mar 17;100(6):693-702. doi: 10.1016/s0092-8674(00)80705-9. PMID 10761934
- [Background] Conneally PM, Dumont-Driscoll M, Huntzinger RS, Nance WE, Jackson CE. Linkage relations of the loci for Kell and phenylthiocarbamide taste sensitivity. Hum Hered. 1976;26(4):267-71. doi: 10.1159/000152813. PMID 976995